CLINICAL TRIAL: NCT01449253
Title: Comparison of Efficacy Different Treatment Regimens in Pulmonary Hypertension Secondary to Lung Disease and or Hypoxia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, S.K.SHARMA, HOD Medicine, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pulmonary hypertension
Record Dates: First submitted 2011-10-07; First posted 2011-10-10 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Pulmonary Hypertension Secondary to Lung Disease and/or Hypoxia
MeSH Terms: interventions — Sildenafil Citrate; Bosentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Monotherapy (Active Comparator): Sildenafil will be started at 20mg OD and then increased to 20mg TDS if there is no fall in BP. Total duration is of 6 months
  Interventions: Drug: Sildenafil
- Sequential Therapy (Active Comparator): Bosentan will be started at 62.5mg BD for 4 weeks and then increased to 125mg BD. Sildenafil will be started be added after 3 months. Sildenafil will be started at 20mg OD and then increased to 20mg TDS if there is no fall in BP. Total duration is of 6 months. Bosentan and sildenafil will be in combination in the last 3 months. No fixed dose combination will be used.
  Interventions: Drug: Sildenafil; Drug: Bosentan
- Combination therapy (Active Comparator): Bosentan will be started at 62.5mg BD for 4 weeks and then increased to 125mg BD. Sildenafil will be started at 20mg OD and then increased to 20mg TDS if there is no fall in BP. Total duration is of 6 months. No fixed dose combination will be used.
  Interventions: Drug: Sildenafil; Drug: Bosentan

INTERVENTIONS:
Drug: Sildenafil — 20 mg initially and then increased to 20 mg TDS if there is no fall in BP
Drug: Bosentan — Bosentan 62.5 mg BD initially for 1 month and then increased to 125 mg BD
  Arms: Combination therapy; Sequential Therapy

SUMMARY:
This is an open label, randomized, interventional study indented to find the efficacy of different treatment regimens in treatment of pulmonary hypertension secondary to lung disease and/or hypoxia.This is to find out when to start combination therapy (sildenafil plus bosentan) in treatment of pulmonary hypertension secondary to lung disease and/or hypoxia.

DETAILED DESCRIPTION:
This is an open label, randomized, interventional study indented to find the efficacy of different treatment regimens in treatment of pulmonary hypertension secondary to lung disease and/or hypoxia. It involves 3 arms, one getting monotherapy with sildenafil for 6 months, 2nd getting bosentan monotherapy initially for 3 months and then combination of sildenafil and bosentan for 3 months, 3rd getting combination sildenafil and bosentan from the beginning for 6 months. The aim is to decide when is the best time to start combination therapy either from start or at the time of drug failure. Improvement will be assessed by change in functional class, pulmonary pressures measured by ECHO, pulmonary function test, six minute walk test and biochemical markers. Lack of randomized trials and Indian data is there on the subject. Also adverse events and serious adverse events will be closely monitored and reported to the ethics committee and DCGI immediately.

ELIGIBILITY:
Inclusion Criteria:

1. Pulmonary artery hypertension diagnosed by doppler echocardiography as mean pulmonary artery pressure 25 mmHg (done in department of cardiology, AIIMS)
2. Age more than 18 years
3. Pulmonary artery hypertension due to hypoxia, either chronic obstructive airway disease or diffuse pulmonary lung disease
4. Willing to consent to participate in the trial
5. WHO functional class I,II, III

Exclusion Criteria:

1. WHO functional class IV
2. Patient participating in any other trial
3. Concomitant coronary artery disease
4. Nitrate intake
5. Liver dysfunction
6. Pregnancy and lactation -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-08; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Echocardiogram | 6 months
  Improvement in pulmonary artery pressures
WHO functional classification | 6 months
  Improvement in WHO functional classification
6 minute walk test | 6 months
  Improvement in 6 minute walk test
Pulmonary function test | 6 months
  Improvement in Pulmonary function test
Visual analog scale for dyspnea | 6 months
  Improvement in Visual analog scale for dyspnea

SECONDARY OUTCOMES:
Echocardiography measuring pulmonary artery pressure | 3 months
  Improvement in pulmonary artery pressures measured by Echocardiography
WHO functional classification | 3 months
  Improvement in WHO functional classification
6 minute walk test | 3 months
  Improvement in 6 minute walk test
Pulmonary function test | 3 months
  Improvement in Pulmonary function test
Visual analog scale for dyspnea | 3 months
  Improvement in Visual analog scale for dyspnea
Biochemical markers at 3 and 6 months | 6 months
  Levels of biomarkers such as Trop T, pro-BNP, uric acid at 3 months and 6 months after starting the drugs
Monitoring side effects of the drugs | 6 months
  adverse events and serious adverse events will be closely monitored and reported to the ethics committee and DCGI immediately

CONTACTS AND LOCATIONS:
Overall Officials: Surendra K. Sharma, MD,Ph.D, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All India Institute Of Medical Sciences, New Delhi, National Capital Territory of Delhi, India